CLINICAL TRIAL: NCT00174837
Title: Phase III Randomized Trial of Concomitant Radiation, Cisplatin, and Tirapazamine Versus Concomitant Radiation and Cisplatin in Patients With Advanced Head and Neck Cancer
Brief Title: TRACE: Tirapazamine-Radiation And Cisplatin Evaluation
Acronym: TRACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC5512; SR259075
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Tirapazamine; Head and Neck Cancer; Cisplatin; Radiation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Tirapazamine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tirapazamine + Cisplatin (Experimental)
  Interventions: Drug: Tirapazamine; Drug: Cisplatin
- Cisplatin (Active Comparator)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Tirapazamine — in combination with cisplatin and concomitant radiation
  Other Names: SR259075
  Arms: Tirapazamine + Cisplatin
Drug: Cisplatin — with concomitant radiation

SUMMARY:
The trial will compare the efficacy and safety of concomitant chemoradiation with tirapazamine, cisplatin and radiation versus cisplatin and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
* Stage III or IV disease (excluding T1N1, and T2N1 and metastatic disease).
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Absolute neutrophil count at least 1.5 X 10^9/L, platelet count at least 100 X 10^9/L, and hemoglobin > 9g/dL.
* Serum bilirubin < 1.25 times upper limit of normal (ULN) and aspartate aminotransferase (AST)/alanine transaminase (ALT) < 2.5 times ULN.
* Calculated creatinine clearance (Cockcroft-Gault) > 55 mL/min.

Exclusion Criteria:

* Metastatic Disease
* Primary cancers of the nasal and paranasal cavities and of the nasopharynx
* Significant intercurrent illness that will interfere with the Chemotherapy or Radiation Therapy during the trial
* Symptomatic peripheral neuropathy > grade 2
* Clinically significant hearing impairment
* Significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Study period

SECONDARY OUTCOMES:
Failure Free Survival, Time To Loco-Regional Failure, Patterns of Failure | Study period
Initial Response Rates at 2 Months After Completion of Chemoradiation Therapy, Final complete response (CR) Rate at Six Months After Completion of Therapy | Study period
Change in QoL From Baseline, Percent of Patients Who Are Feeding Tube Dependent 12 Months After Completion of Therapy | Study period
Toxicity and Safety | Study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- sanofi-aventis New Zealand administrative office, Macquarie Park, New Zealand
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com